CLINICAL TRIAL: NCT02288078
Title: A Study of Prophylactic Oral Steroids for Fatigue and Malaise Due to Regorafenib Treatment for Unresectable Metastatic Colorectal Cancer: a Randomized, Placebo-controlled, Double-blind Phase 2 Clinical Study (KSCC1402/HGCSG1402)
Brief Title: Oral Steroids for Regorafenib-induced Fatigue/Malaise in Unresectable mCRC (KSCC1402/HGCSG1402)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Research Support Center Kyush (Other)
Responsible Party: Principal Investigator, Hideo Baba, Professor, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KSCC1402/HGCSG1402; UMIN000015131 (Registry Identifier: University Hospital Information Network)
Record Dates: First submitted 2014-10-28; First posted 2014-11-11 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Rectal Cancer
Keywords: unresectable colorectal cancer; regorafenib; Steroid; fatigue and malaise; Phase 2 randomized, controlled trial (RCT)
MeSH Terms: conditions — Rectal Neoplasms; Fatigue | interventions — Blood Pressure; Patient Reported Outcome Measures; Hematologic Tests; Blood Chemical Analysis; Blood Coagulation; Urinalysis; Dexamethasone; regorafenib; Proton Pump Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Active Comparator): Treatment with regorafenib (160 mg/day, oral administration, 3 weeks on therapy followed by 1 week off therapy), test drug capsule (dexamethasone 2 mg) and proton pump inhibitors (PPIs) will be started within 14 days of enrollment. The protocol treatment period is 4 weeks.
  Follow-up treatment for the underlying disease after the 4-week protocol treatment is not specified. The physician in charge will decide whether or not to continue treatment with regorafenib. For the prevention of fatigue/malaise, dexamethasone 2 mg can be used.
  General condition, blood pressure, Patient Reported Outcome, clinical findings, hematology/blood chemistry, coagulation and fibrinolysis system, urinalysis, medicatiob check, adverse event, thyroid function test, brain MRI, Contrast-enhanced torso CT
  Interventions: Other: General condition; Other: Blood pressure; Other: Patient Reported Outcome; Other: Clinical findings; Other: Hematology/blood chemistry; Other: Coagulation and fibrinolysis system; Other: Urinalysis; Other: Medication check; Other: Adverse event; Other: Thyroid function test; Other: Contrast-enhanced torso CT; Other: Brain MRI; Drug: Dexamethasone; Drug: Regorafenib; Drug: Proton pump inhibitor
- Placebo group (Placebo Comparator): Treatment with regorafenib (160 mg/day, oral administration, 3 weeks on therapy followed by 1 week off therapy), placebo capsule (lactose) and proton pump inhibitors (PPIs) will be started within 14 days of enrollment. The protocol treatment period is 4 weeks.
  Follow-up treatment for the underlying disease after the 4-week protocol treatment is not specified. The physician in charge will decide whether or not to continue treatment with regorafenib. For the prevention of fatigue/malaise, dexamethasone 2 mg can be used.
  General condition, blood pressure, Patient Reported Outcome, clinical findings, hematology/blood chemistry, coagulation and fibrinolysis system, urinalysis, medication check, adverse event, thyroid function test, brain MRI, Contrast-enhanced torso CT
  Interventions: Other: General condition; Other: Blood pressure; Other: Patient Reported Outcome; Other: Clinical findings; Other: Hematology/blood chemistry; Other: Coagulation and fibrinolysis system; Other: Urinalysis; Other: Medication check; Other: Adverse event; Other: Thyroid function test; Other: Contrast-enhanced torso CT; Other: Brain MRI; Drug: Regorafenib; Drug: Placebo; Drug: Proton pump inhibitor

INTERVENTIONS:
Other: General condition — Eastern Cooperative Oncology Group (ECOG) performance status (PS), height and body weight
Other: Blood pressure — systolic blood pressure (SBP)/diastolic blood pressure (DBP)
Other: Patient Reported Outcome — Incidence of fatigue or malaise (All grade of CTCAE ver. 4), anorexia, Brief fatigue inventory (BFI), FACT-C.
  Other Names: PRO
Other: Clinical findings — * Blood and lymphatic system disorders: febrile neutropenia
  * Gastrointestinal disorders: constipation, diarrhea, oral mucositis, nausea, and vomiting
  * General disorders and administration site conditions: fatigue and malaise
  * Immune system disorders: allergic reaction
  * Metabolism and nutrition disorders: anorexia
  * Nervous system disorders: dysgeusia and peripheral sensory neuropathy
  * Respiratory, thoracic and mediastinal disorders: hoarseness (change of voice)
  * Skin and subcutaneous tissue disorders: alopecia, skin hyperpigmentation, urticaria, and palmar-plantar erythrodysesthesia syndrome
  * Vascular disorders: hypertension
  * Symptomatic pancreatitis
Other: Hematology/blood chemistry — White blood cell count, absolute neutrophil count (stab + segmented), hemoglobin, platelet count, albumin, total bilirubin, aspartate aminotransferase(AST) (GOT), alanine aminotransferase (ALT) (GPT), serum creatinine, Na, K
Other: Coagulation and fibrinolysis system — international normalized ratio (INR)
Other: Urinalysis — Proteinuria (qualitative)
Other: Medication check — Medicine taking situation (regorafenib, dexamethasone and placebo) determined by subject's diary at every courses
Other: Adverse event — CTCAE ver.4.0
  Other Names: AE
Other: Thyroid function test — Thyroid-stimulating hormone (TSH), T4, and T3
Other: Contrast-enhanced torso CT — It is recommended that CT images should be taken every 4 weeks (if possible) or at least every 8 weeks (allowable time window: ± 2 weeks), with the treatment phase taken into consideration.
Other: Brain MRI — If any symptom of brain metastasis is suspected
Drug: Dexamethasone — Capsule filled with dexamethasone and lactose
  Other Names: DX
  Arms: Treatment group
Drug: Regorafenib — Film-coating tablet contains 40 mg of regorafenib
  Other Names: Stivarga
Drug: Placebo — Capsule filled with lactose
  Other Names: PL
  Arms: Placebo group
Drug: Proton pump inhibitor — PPIs (omeprazole, lansoprazole, etc, as not specified) for prevention of peptic ulcer
  Other Names: PPI

SUMMARY:
The objective of this randomized placebo-controlled Phase 2 study is to evaluate prophylactic effects of dexamethasone for fatigue and malaise (weakness, lethargy, malaise) resulting from regorafenib treatment, as well as to assess treatment continuation of regorafenib.

DETAILED DESCRIPTION:
1. Patient registration procedure

   If it is confirmed that the subject meets the inclusion criteria and correspondent none of the exclusion criteria, the subject is registered by using Clinical Research Support Center (CReS) Kyushu registration/allocation system. The registration with the registration/allocation system is available for 24 hr (URL: https://reg.cres-kyushu.or.jp/qmin/login/) and needs for individual identifier (ID) and password.
2. Quality management

   * Preparation and management of the test drugs

The test drugs are an active drug, which is a capsule filled with dexamethasone powder and lactose, and a placebo, which is a capsule filled with only lactose. The test drugs will be prepared by the Department of Pharmacy (manager: Professor Masuda), Kyushu University Hospital in accordance with the procedures for preparation of the test drugs. Dexamethasone powder and lactose will be purchased by Department of Surgery and Science, Graduate School of Medical Sciences, Kyushu University from Tomita Pharmaceutical and delivered to the pharmacy department. Research funds will be used for the purchase. The capsule will be purchased from Tomita Pharmaceutical. The test drugs will be delivered to CReS-Kyushu (enrollment/data center) and managed using a double-blind method in accordance with the procedures. The double-blind code will be kept by the person responsible for management of the test drugs Shoji Tokunaga, Medical Information Center, Kyushu University, and a backup of the code will be kept by Hidekazu Aratani of CReS-Kyushu.

The test drugs will be managed according to the investigational drug number and stored at the warehouse of the Fukuoka branch of Yamato Logistics Co., Ltd. The warehouse is certified to store drugs for humans for more than 2 years under the supervision of pharmacists.

In the participating medical institution, manager and vice manager for the management of the test drugs will be appointed. It is preferable that the manager and vice managers are selected from among personnel who are experienced in drug management including personnel from the Department of Pharmacy or clinical trial management office. The manager is not allowed to become the investigator or sub-investigator. A physician who may treat subjects is not allowed to become the manager.

The electronic data capture (EDC) system will be used for communications between the enrollment/data center, Yamato Logistics and participating medical institution. Information on subjects will be reported by e-mail to the data center, and the data center will ensure the information by telephone to Yamato Logistics and the investigational drug management division of the medical institution. The test drugs will be delivered by Yamato Logistics to the medical institution. The test drugs for only a subject will be delivered once (allocation adjustment factor). Considering that a number of days are necessary for delivery, there should be at least 3 working days between enrollment and start of treatment. The interval between enrollment and start of treatments should be up to 14 days. Physicians treating subjects are not allowed to manage the test drugs. The vice manager will manage the test drugs according to subjects under the supervision of the manager. Orders for the test drugs will be made by letter or e-mail in accordance with the medical institution's procedures. A sufficient number of capsules of the test drugs until the next hospital visit will be ordered/prescribed once. If the test drugs are used properly in accordance with the protocol, an order/prescription for the test drugs will be made every 7 days. Subjects (patients) will be advised to keep records of the use of regorafenib and test drugs in the medication diary. The remaining number of capsules of the test drugs will be checked in consideration of the use of the test drugs. The remaining test drugs will be returned to the study office. In accordance with the protocol, the test drugs should be prescribed for 28-day treatment, but will be prescribed for 30-day treatment considering loss and damage. The test drug for 2-day treatment should be left unused when treatment is completed. The remaining test drugs will be returned to the enrollment/data center.

When the test drugs are delivered, the enrollment number, investigational drug number, reception date, the number of capsules of the test drugs delivered will be entered in the EDC system. Also, the number of capsules prescribed, date of prescription, remaining number of capsules (total number of capsules stored including the number of capsules returned), confirmation date of completion/discontinuation of the protocol treatment, total remaining number of capsules including the number of capsules returned will be entered in the EDC system.

The number of capsules lost and reasons for the loss will be entered in the EDC system.

* Monitoring

A central monitoring or in-site monitoring are carried out based on the data from case report form (CRF) collecting at data coordinating center. In principle, an on-site monitoring is not carried out, but it may be carried out when the on-site monitoring is determined to need by Kyushu Study group of Clinical Cancer (KSCC) steering committee from the results of the central monitoring so on.

Data Monitoring Committee A Data Monitoring Committee (DMC) has been established.

* Data entry

all data will be entered by the double entry method. Referential data rules, valid values, range checks, and consistency checks against data already stored in the database will be supported. Checks will be applied at the time of data entry into a specific field. Additional errors will be detected by programs designed to detect missing data or specific errors in the data. The investigator who receives the inquiry will respond by checking the original forms for inconsistency, checking other sources to determine the correction, modifying the original paper form entering a response to the query.

* Regular monitoring report

A regular monitoring report generated by data coordinating center is submitted to KSCC Steering Committee, principal investigator, the DMC etc and it is reviewed according to "KSCC regulation on the monitoring". The information on the status of site ethics committee (EC) approval and the achievement of enrollment: number of enrollment- total/per periodical, total/per site, is reported monthly using e-mail.

* Contents of monitoring report

Study abstract: schema/purpose/subject/endpoint/definition of treatment/anticipated enrollment number/progress of the study Enrollment status: per participating site/total Monitoring activity: contents of activity/CRF collection per site/uncollected CRF, inquiry Review of the eligible treatment case：the case of ineligible possibility/the case determined as ineligible/number of eligible case/the case determined as non-treatment/total number of treatment case Review of a target population for analysis: the number of cases targeted for efficacy analysis/safety analysis Patient background Treatment time-course: summary of on-treatment and discontinuation/summary of reason for discontinuation/list of reason for discontinuation Protocol violation/deviation Safety evaluation: serious adverse reaction, event/the case which was notified to the study group among the adverse reactions, events with an ordinary report/general adverse events Others

* Audit

A site audit is carried out by the audit members of KSCC Coordinating Center, data coordinating center, medical staff of other site under the approval of the site director according to "KSCC regulation for site audit". The results of the audit are reported to the site director, KSCC Steering Committee, principal investigator etc. (if required, to DMC).

ELIGIBILITY:
Inclusion Criteria:

* Capable of granting informed consent in writing for receiving treatment outlined in this protocol
* The investigators determines that the patient can receive the treatment outlined in this protocol
* Histological diagnosis of adenocarcinoma of either the colon or the rectum, regardless of RAS mutation
* Metastatic colorectal cancer scheduled for treatment with regorafenib
* Lesions are either measurable or non-measurable according to RECIST ver. 1.1
* Contrasted torso CT within 28 days before enrollment
* At least 20 years of age
* PS 0-1
* Bone marrow, hepatic, and renal functions have all been confirmed as normal within 14 days prior to initiation of regorafenib treatment
* Life expectancy of at least 3 months

Exclusion Criteria:

* Used regorafenib previously
* Blood transfusion or granulocyte-colony stimulating factor (G-CSF) administration within 14 days
* Grade 2 or higher fatigue or malaise or asthenia according to NCI-CTCAE ver. 4.0
* History of a different type of cancer according to histological findings or cancer of a different primary focus within the past 5 years. The following are excluded: carcinoma in situ of the cervix, non-melanoma skin cancer, superficial bladder cancer (Ta, Tis, and T1), gastric cancer,non-invasive breast cancer, etc
* Highly invasive surgery, an open biopsy, or who have received significant trauma within 28 days of initiating regorafenib treatment
* Congestive cardiac failure of New York Heart Association (NYHA) >=Class 2
* Unstable angina (symptoms at rest),new-onset angina (onset within past 3 months), or a history of myocardial infarction within 6 months of initiating treatment
* Arrhythmia requiring treatment with anti-arrhythmia drugs
* Uncontrollable hypertension
* Pleural effusion or ascites causing dyspnea (NCI-CTCAE >=Grade 2)
* History of venous or arterial thrombosis or embolism within 6 months prior to initiation of treatment, including cerebrovascular accidents, deep vein thrombosis, or pulmonary embolism
* Patients with active infections of NCI-CTCAE >=Grade 3
* Positive for either hepatitis B (HB)s antigen or hepatitis C virus (HCV) antibody
* Seizure disorders requiring drug treatment
* Cerebral metastases or history of such
* History of organ transplant
* Symptoms or history of hemorrhagic tendency, regardless of severity
* Some form of hemorrhaging (NCI-CTCAE >=Grade 2) within 4 weeks prior to initiating treatment
* Incurable wound, fracture or ulcer
* Renal failure requiring either hemodialysis or peritoneal dialysis
* Dehydration symptoms of NCI-CTCAE >=Grade 1
* Abusing drugs or who are in a physical, psychological, or social state which might impair study participation or evaluation of results
* Interstitial lung disease with active signs or symptoms
* Have difficulty taking oral drugs
* Digestion absorption disorders
* Adverse events resulting from previous treatments or procedures which have not yet resolved (NCI-CTCAE >=Grade 2)
* Received systemic anti-cancer treatments within 2 weeks prior to initiation of regorafenib treatment, including chemotherapy, molecular target drugs, immunotherapy, or hormone therapy
* Poorly controlled glucose tolerance abnormalities due to diabetes mellitus (patients using insulin)
* Active GI ulcers or a history of such
* Glaucoma
* Oral steroids are otherwise contraindicated
* Either pregnant or nursing. Women who may become pregnant must have a negative pregnancy test within 7 days prior to initiating treatment
* Women who may become pregnant, or men whose partners may become pregnant, must agree to use appropriate contraceptives from granting of consent to 3 months after conclusion of regorafenib therapy
* Other illnesses or conditions which, according to the judgment of the investigator, may result in physical harm caused by the study, or which may impair study compliance

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
incidence of fatigue or malaise (CTCAE ver. 4, all grades) | 4weeks
  With the number of subjects in safety analysis set (SAS) as the denominator, the frequency of the worst grade of "fatigue" or "malaise"(according to CTCAE ver.4.0) is determined.

SECONDARY OUTCOMES:
brief fatigue inventory （Patient Reported Outcome） | 4weeks
  For all subjects enrolled in the present clinical study, the severity of fatigue/malaise is rated using the brief fatigue inventory (BFI) scale obtained every week following the start. Mean of numerical evaluating scale from 9 questions is defined as the global fatigue score. Details of the method to collect and analyze the BFI as a patient reported outcome (PRO) will be specified in a procedure separately prepared along the instruction by Professor Yamaguchi (Tohoku University).
adverse events | 1year
  With the number of subjects in whom at least a part of the protocol treatment is provided (all treated subjects) set as the denominator, the frequencies of the following adverse events/toxicity (according to CTCAE ver.4.0) appearing at the worst grade whenever during the entire treatment course are determined by treatment group. Whether ineligible subjects are included in the analysis set or not is decided by the KSCC's research administration office through discussion with the Registration/Data Center.
  With the number of subjects in Full analysis set (FAS) set as the denominator, the rate of treatment discontinuation due to adverse events other than disease progression is determined.
relative dose intensity (regorafenib) | 4weeks
  With the planned dose of regorafenib in 1 course set as the denominator while the actual dose set as the numerator, the relative dose intensity (given in percentage) is determined for the FAS.

OTHER OUTCOMES:
medicine taking situation (regorafenib, study drug) | 4weeks (study drug), 1year (regorafenib)
response rate | 1year
  The best response rate based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 is defined as the proportion of subjects (among the FAS) whose best overall response is either complete response (CR) or partial response (PR).
disease control rate (DCR) | 1year
  The disease control rate is defined as the proportion of subjects (among the FAS) whose best overall response and confirmed overall response based on RECIST v1.1 are either of CR, PR, or stable disease (SD).
treatment continuation period | 1year
progression-free survival (PFS) | 1year
  For the FAS, the progression-free survival is defined as a period from the day of enrollment to whichever earlier date of exacerbation or death from any cause.
overall survival (OS) | 1year
  Taking the enrollment day as the starting date, the overall survival is defined as time to death for any cause.
  Subjects who are alive are censored for over survival at the date that they are last known to be alive.
  Subjects who lost to follow-up are censored for overall survival at the date that they are last known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Yasunori Emi, MD, PhD, Study Director — Saiseikai Fukuoka General Hospital
Locations (1):
- Saiseikai Fukuoka General Hospital, Fukuoka, Japan